CLINICAL TRIAL: NCT03362398
Title: LC-MS/MS Quantitative Determination of Omarigliptin & Trelagliptin in Twelve Healthy Egyptian Volunteers' Plasma
Brief Title: Omarigliptin & Trelagliptin in Twelve Healthy Egyptian Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Bassam Mahfouz Ayoub, Lecturer of Chemistry, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CDRD-4
Record Dates: First submitted 2017-11-20; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; trelagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omarigliptin (Active Comparator): Drug: Omarigliptin 25 mg
  Interventions: Drug: Omarigliptin 25 mg
- Trelagliptin (Active Comparator): Drug: Trelagliptin 100 mg
  Interventions: Drug: Trelagliptin 100 mg

INTERVENTIONS:
Drug: Omarigliptin 25 mg — Once weekly new anti-diabetic drug approved only in Japan
  Other Names: Zafatek tablets
  Arms: Omarigliptin
Drug: Trelagliptin 100 mg — Once weekly new anti-diabetic drug approved only in Japan
  Other Names: Marizev tablets
  Arms: Trelagliptin

SUMMARY:
The proposed study will consider the LC-MS/MS quantitative determination of Omarigliptin & Trelagliptin after administration to twelve Egyptian volunteers. The main aim of the study is to confirm that the developed LC-MS/MS method is applicable for the bio-assay of the drugs in the actual biological samples at the time of Cmax (nearly about 1.5 hours). The design of the study is open labeled, randomized, one treatment, one period, single dose study. The concentration of the drugs after 1.5 h will be determined in healthy human subjects according to the ethical regulations of World Medical Association Declaration of Helsinki (October 1996) and the International Conference of Harmonisation Tripartite Guideline for Good Clinical Practice. Written informed consent was provided (attached and signed by the twelve volunteers) in order to be approved by the ethics committee of the Faculty of Pharmacy, The British University in Egypt. The good health of the human subjects was confirmed by a complete medical history and physical examination. Samples from twelve, healthy, adult, male, smoking, Egyptian volunteers (age: 23-37 years, Average weight: 81.6 kg, Average BMI: 30.4) will be collected at 1.5 h, to be transferred to heparinized centrifuge tubes in order to be analyzed by LC-MS/MS study (developed & validated) after single oral dose administration of one Marizev® tablet nominally containing 25 mg of Omarigliptin (first arm as 6 volunteers) or one Zafatek® tablet nominally containing 100 mg of Trelagliptin (second arm as 6 volunteers). The blood samples (0.5 mL of each sample) will be centrifuged at 3000 rpm for 5 minutes, 100 µL of the plasma will be separated and spiked with the internal standard working solution and then the sample preparation and LC-MS/MS determination will be applied. Blood glucose level will be determined for all volunteers at different time intervals to monitor any hypoglycemic effect to ensure their safety all over the study. The study will be conducted as per FDA guidelines & the evaluation of safety of the study will be based on monitoring of blood glucose level, vital signs, pulse rate, monitoring of adverse events, and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Must be able to swallow tablets

Exclusion Criteria:

* Insulin dependent diabetes
* Type-2 diabetes
* Hospitalized within 1 week

Ages: 23 Years to 37 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Human plasma concentration of 12 participants will be measured after 1.5 h | 2 weeks
  The main purpose of this outcome is to check the suitability of the developed LC-MS/MS method for determination of the drugs in human plasma

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Egypt